CLINICAL TRIAL: NCT00744302
Title: Study of 1.25 mmol/L Calcium Dialysate on Mineral Metabolism in Haemodialysis Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGHD-001
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Hyperparathyroidism; Hypercalcemia
Keywords: Dialysate calcium; Mineral metabolism; Parathyroid hormone; Calcification; Cardiovascular disease; Haemodialysis
MeSH Terms: conditions — Hyperparathyroidism; Hypercalcemia; Calcinosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCD (Experimental): Physiological calcium (1.25 mmol/L) dialysate therapy All subjects in the study phase will continue to take calcium carbonate and/or active vitamin D agents.
  Interventions: Drug: physiological (1.25 mmol/L ) calcium dialysate
- NCD (Active Comparator): Normal calcium (1.5 mmol/L) dialysate therapy All subjects in the study phase will continue to take calcium carbonate and/or active vitamin D agents.
  Interventions: Drug: physiological (1.25 mmol/L ) calcium dialysate

INTERVENTIONS:
Drug: physiological (1.25 mmol/L ) calcium dialysate — Using the physiological calcium dialysate (1.25 mmol/L calcium dialysate)for Stable haemodialysis treatment for more than 3 months, undergoing 2 to 3 times haemodialysis a week for 4 to 5 hours per session

SUMMARY:
A prospective, randomized, controlled multicenter trial to evaluate 1.25 mmol/L (physiological) vs. 1.5 mmol/L calcium dialysate on serum markers of mineral metabolism, secondary hyperparathyroidism and cardiovascular calcification in prevalent haemodialysis patients. And the long term safety of the 1.25 mmol/L calcium dialysate was also considered.

There are two phases of study for each subject. Phase 1 (screening phase). During this phase, each potential subject will be evaluated to determine if he/she is eligible for the study.

Phase 2 (intervention phase). Each subject will be randomly allocated to physiological calcium dialysate (1.25 mmol/L calcium dialysate) group (PCD group), and normal calcium dialysate (1.5 mmol/L calcium dialysate) group (NCD group). The follow-up duration was 36 months.

DETAILED DESCRIPTION:
All patients recruited from these centers who met the inclusion criteria were randomly allocated to physiological calcium dialysate (1.25 mmol/L calcium dialysate) group (PCD group), and normal calcium dialysate (1.5 mmol/L calcium dialysate) group (NCD group). The follow-up duration was 36 months.

Calcium carbonate was mainly used as the phosphate binder. Active vitamin D metabolite, calcitriol (Rocaltrol, Hoffmann La Roche, and Basel, Switzerland) was given as to control the secondary hyperparathyroidism. The doses of these agents were adjusted according to the serum calcium level, serum phosphate level, calcium-phosphorus product and serum iPTH level, which were recommended by the K/DOQI Guidelines 6.3b and 8B. Aluminum hydroxide might be introduced as a phosphate binder for no more than 4 weeks in addition to calcium carbonate and dietary restriction when serum phosphate level could not get a good control (serum P level≥1.78 mmol/L, lasting above 4 weeks). A non- calcium-containing phosphate binder could be administered for 1~2 weeks in patients with hypercalcaemia during the observation. At the time of the study, non-calcium, non-aluminum based phosphate binders as well as calcium acetate were not available in our country.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Stable haemodialysis treatment for more than 3 months, undergoing 2 to 3 times haemodialysis a week for 4 to 5 hours per session
* Secondary hyperparathyroidism defined as serum intact parathyroid hormone (iPTH) > 150 pg/mL, hypercalcemia defined as serum Ca > 2.2 mmol/L and /or calcium phosphate product ≥55mg2/dl2

Exclusion Criteria:

* Inability or unwillingness to sign the informed consent
* Cardiac arrhythmia
* Serious renal osteopathy
* Oral active vitamin D and/or calcium carbonate intolerance
* Poor compliance or unwillingness to meet the scheme demands raised by the investigators
* Patients who had undergone percutaneous ethanol injection therapy or parathyroidectomy for secondary hyperparathyroidism
* Patients who had previously been treated and/or were being treated with glucocorticoid, which affects bone metabolism.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2006-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Improvement of mineral metabolism and remission of secondary hyperparathyroidism | 2006-2009

SECONDARY OUTCOMES:
Improvement of cardiovascular calcification and decrease of clinical cardiovascular events | 2006-2009

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University; Tanqi Luo, MD, Principal Investigator — Department of Nephrology, 3rd Affiliated Hospital of Sun Yet-Sen University; Qiong Luo, MD, Principal Investigator — Department of Nephrology, Shen Zhen Affiliated Hospital of Peking University; Yaozhong Kong, MD, Principal Investigator — Department of Nephrology, the 1st People's Hospital Fo Shan City; Wei Shi, MD, Principal Investigator — Department of nephrology, People's Hospital of Guangdong Province; Haitang Hu, MD, Principal Investigator — Department of Nephrology, People's Hospital Shun De City; Zaiseng Zhou, MD, Principal Investigator — Department of Nephrology, People's Hospital of Zhongshan City
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China